CLINICAL TRIAL: NCT02704208
Title: A Technology-Delivered Peer-to-Peer Support ART Adherence Intervention for Substance-using HIV+ Adults
Acronym: TWM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); Center for HIV Educational Studies & Training (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1504S69721; 1R01DA039950-01 (NIH)
Record Dates: First submitted 2016-03-04; First posted 2016-03-09 (Estimated); Results first posted 2023-06-07 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-06

CONDITIONS: HIV
Keywords: Antiretroviral Therapy; Medication Adherence; Technology-based Intervention
MeSH Terms: conditions — Medication Adherence | interventions — Nicotine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Behavioral: Thrive With Me Intervention (Experimental): Participants randomized to the TWM Intervention will gain access to a website for 150 days. The TWM website includes: peer-to-peer support through a private social network and optimized gaming features; daily SMS communication for medication reminders and mood tracking; medication adherence monitoring; and tailored HIV informational content.
  Interventions: Behavioral: Thrive With Me Intervention
- Behavioral: Thrive With Me Control (Placebo Comparator): Participants randomized to the TWM Control group will receive HIV related content through a weekly web link. The web links will be static pages (not interactive) with information aimed at improving overall wellbeing while living with HIV, but not focused on improving ART medication adherence.
  Interventions: Behavioral: Thrive With Me Control

INTERVENTIONS:
Behavioral: Thrive With Me Control — Those assigned to the TWM control group will receive a weekly email with static HIV informational content. Information will be focused more on quality of life and general wellbeing issues and will not be specific to medication adherence.
  Other Names: TWM Control
  Arms: Behavioral: Thrive With Me Control
Behavioral: Thrive With Me Intervention — Those assigned to the TWM intervention will have 150 days to access tailored content on a mobile-enhanced website. They will also have social support through a network of other HIV-positive men. Finally they will track their daily ART medication adherence and mood through SMS and website use.
  Other Names: TWM Intervention
  Arms: Behavioral: Thrive With Me Intervention

SUMMARY:
The "Thrive With Me" (TWM) trial is testing the efficacy of a mobile enhanced website aimed at improving Antiretroviral Therapy (ART) adherence for HIV-positive men who have sex with men (MSM). TWM is a technology-delivered peer-to-peer social support intervention with social networking and gaming components. In addition to real-time peer-to-peer support capabilities, the TWM intervention provides participants with Antiretroviral Therapy (ART) adherence self-monitoring tools, medication dose reminders, and HIV-related informational content.

DETAILED DESCRIPTION:
The "Thrive with Me" (TWM) intervention is a technology-delivered peer-to-peer social support intervention grounded in the Information, Motivation, and Behavioral Skills (IMB) model for HIV positive men who have sex with men (MSM). In addition to asynchronous peer-to-peer support capabilities, the TWM intervention provides participants with Antiretroviral Therapy (ART) adherence self-monitoring tools, medication dose reminders, and HIV-related informational content. Based on the encouraging findings of the TWM pilot study (completed in 2011) and the need for novel, evidence-based effective ART adherence interventions, we propose the following study aims for this full-scale RCT. Primary aims (Aims 1 and 2) are to examine the efficacy of the online and mobile-enabled TWM intervention in a full-scale randomized controlled trial. HIVpositive adults (all men who have sex with men [MSM]) with detectable HIV viral load (VL) residing in New York City will be randomized to receive the TWM intervention or an information-only HIV/ART intervention for a 6-month period. Recruitment will be stratified by recent drug use, such that half will report recent illicit drug use. HIV VL, validated self-reported ART adherence, and intervention utilization measures will be collected at baseline, post-intervention, and 6-, and 12- month follow up. We hypothesize that participants in the TWM intervention will demonstrate significant improvements in self-reported ART adherence and VL at each follow-up time point compared to control participants, with greatest improvements among recent drug users. Aim 3 (a secondary aim) is to examine the effects of the intervention on theory-based change processes (i.e., IMB factors and social support) for improving VL, ART adherence, and substance use outcomes. We hypothesize that tailored adherence information, motivation for adherence, adherence behavioral skills, and peer social support will be associated with VL suppression and improved ART adherence and drug use outcomes. All study participants will reside in the New York City metropolitan area. The Center for HIV Education Studies and Training at CUNY Hunter College is overseeing the recruitment, enrollment, and retention of human subjects. The primary outcome measure is biological viral load (VL) at each assessment period. Specifically, blood draws will be taken at baseline, immediate post-intervention, 6- and 12-month post-intervention follow-up assessment points to assess the effects of the TWM intervention on VL, the most important biological marker for adherence. Plasma VL is considered undetectable at <20 copies/mm3 and we will provide test results to participants after each visit. The University of Minnesota IRB is overseeing all human subjects protocols for the study. Brief Summary The "Thrive with Me" (TWM) intervention is a technology-delivered peer-to-peer social support intervention grounded in the Information, Motivation, and Behavioral Skills (IMB) model for HIV positive men who have sex with men (MSM). In addition to asynchronous peer-to-peer support capabilities, the TWM intervention provides participants with Antiretroviral Therapy (ART) adherence self-monitoring tools, medication dose reminders, and HIV-related informational content. This is a randomized control efficacy trial of the TWM intervention. The primary outcome measure is biological viral load (VL) at each assessment period. All study participants will reside in the New York City metropolitan area. The Center for HIV Education Studies and Training at CUNY Hunter College is overseeing the recruitment, enrollment, and retention of human subjects.

ELIGIBILITY:
Inclusion Criteria:

1. 18+ years of age;
2. Male gender;
3. Sex with 1+ men in the prior year;
4. Diagnosis of HIV and currently prescribed ART;
5. Self-reported detectable VL in past 12 months OR self-reported problems with HIV medication adherence;
6. Residing in the New York City metropolitan area and availability meet with project staff at each assessment time point; and
7. English-speaking (since the intervention will be in English).
8. Self-reported recent drug use (the sample will be stratified by recent drug use and non-recent drug use)

Exclusion Criteria:

1. 17 years of age or younger;
2. Not male gender;
3. 0 male sex partners in the prior year;
4. No diagnosis of HIV and/or not currently prescribed ART;
5. No self-reported detectable VL in past 12 months OR self- reported very good/excellent HIV medication adherence;
6. Residing outside of the New York City metropolitan area and/or no availability meet with project staff at each assessment time point; and
7. Non-English-speaking (since the intervention will be in English).

Ages: 18 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 410 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Center for HIV Education Studies and Training, Hunter College, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Horvath KJ, Lammert S, Erickson D, Amico KR, Talan AJ, Shalhav O, Sun CJ, Rendina HJ. A Web-Based Antiretroviral Therapy Adherence Intervention (Thrive With Me) in a Community-Recruited Sample of Sexual Minority Men Living With HIV: Results of a Randomized Controlled Study. J Med Internet Res. 2024 Sep 30;26:e53819. doi: 10.2196/53819. PMID 39348677
- [Derived] Horvath KJ, Amico KR, Erickson D, Ecklund AM, Martinka A, DeWitt J, McLaughlin J, Parsons JT. Thrive With Me: Protocol for a Randomized Controlled Trial to Test a Peer Support Intervention to Improve Antiretroviral Therapy Adherence Among Men Who Have Sex With Men. JMIR Res Protoc. 2018 May 31;7(5):e10182. doi: 10.2196/10182. PMID 29853437

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Men residing in the New York City metro area were recruited by study staff using active (e.g., direct outreach) and passive (e.g., advertising in clinic settings, internet-based) recruitment approaches. Internet-recruitment efforts were using online venues that cater to the study population and field-based recruitment strategies include conduct on-site preliminary screening via tablets at local bars, clubs, and community events.
Groups:
- Behavioral: Thrive With Me Intervention: Participants randomized to the TWM Intervention gained access to the TWM website for 150 days. The TWM website includes: peer-to-peer support through a private social network and optimized gaming features; daily SMS communication for medication reminders and mood tracking; medication adherence monitoring; and tailored HIV informational content.
- Behavioral: Control Arm: Participants randomized to the TWM Control group will receive HIV related content through a weekly web link. The web links will be static pages (not interactive) with information aimed at improving overall wellbeing while living with HIV, but not focused on improving ART medication adherence.
Period: Overall Study
Arm/Group | Behavioral: Thrive With Me Intervention | Behavioral: Control Arm
Started | 202 | 199
Completed | 160 | 162
Not Completed | 42 | 37
Not completed — Lost to Follow-up | 42 | 37

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Behavioral: Thrive With Me Intervention | Behavioral: Control Arm | Total
Number analyzed (Participants) | 202 | 199 | 401
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.1 (10.8) | 38.1 (10.6) | 39.1 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 202 | 199 | 401
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 62 | 46 | 108
  Not Hispanic or Latino | 140 | 153 | 293
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 4 | 5
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 2
  Black or African American | 123 | 107 | 230
  White | 54 | 59 | 113
  More than one race | 12 | 19 | 31
  Unknown or Not Reported | 9 | 8 | 17
Region of Enrollment [Number; unit: participants]
  United States | 202 | 199 | 401

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants With an Undetectable HIV Viral Load
Description: Undetectable viral load (plasma viral load is considered undetectable at <20 copies/mm3)
Time Frame: up to 17 months period
Measure: Count of Participants; unit: Participants
Arm/Group | Behavioral: Thrive With Me Intervention | Behavioral: Control Arm
Number analyzed (Participants) | 202 | 199
Participants | 107 | 113

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for 17 months (i.e., from baseline to the end of study participation).
Arm/Group | Behavioral: Thrive With Me Intervention | Behavioral: Control Arm
All-Cause Mortality (participants affected / at risk) | 1/202 | 0/199
Serious Adverse Events (participants affected / at risk) | 0/202 | 0/199
Other Adverse Events (participants affected / at risk) | 2/202 | 0/199
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Behavioral: Thrive With Me Intervention (N=202) | Behavioral: Control Arm (N=199)
Suicidal Ideation (Psychiatric disorders) | 2 (3) | 0 (0) — 2 participants expressed suicidal ideation during the course of the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-04-02): https://cdn.clinicaltrials.gov/large-docs/08/NCT02704208/Prot_000.pdf
  • Statistical Analysis Plan (2022-04-29): https://cdn.clinicaltrials.gov/large-docs/08/NCT02704208/SAP_001.pdf